CLINICAL TRIAL: NCT01683838
Title: Double-Blind, Placebo-Controlled, 12-Week Parallel Group Study to Evaluate Safety and Efficacy of Oral Fampridine-SR in Subjects With Moderate to Severe Spasticity Resulting From Chronic, Incomplete Spinal Cord Injury
Brief Title: Safety and Efficacy of Oral Fampridine-Sustained Release (SR) for the Treatment of Spasticity Resulting From Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-F302
Record Dates: First submitted 2012-08-24; First posted 2012-09-12 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2014-01

CONDITIONS: Spinal Cord Injury; Muscle Spasticity
Keywords: spinal cord injury; muscle spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fampridine-SR 50mg/day (Active Comparator)
  Interventions: Drug: Fampridine-SR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fampridine-SR — 25mg bid (twice daily)
  Arms: fampridine-SR 50mg/day
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with spinal cord injury, some fibers may be destroyed at the site of injury, while others remain connected but do not work correctly to carry electrical impulses. As a result, subjects with an incomplete spinal cord injury may have spasticity which is muscle spasms or muscle stiffness that makes movement difficult. Fampridine-SR is an experimental drug that increases the ability of the nerve to conduct electrical impulses. This study will examine the effects of Fampridine-SR on moderate to severe lower-limb spasticity, as well as the effects on bodily functions such as bladder control, bowel function and sexual function. The study will also examine the possible risks of taking Fampridine-SR.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete traumatic Spinal Cord Injury (at least 18 months prior and stable for 6 months)
* Moderate to severe lower-limb spasticity
* Able to give informed consent and willing to comply with protocol

Exclusion Criteria:

* Pregnancy
* History of seizures
* Existing or history of frequent Urinary Tract Infections
* History of drug or alcohol abuse
* Allergy to pyridine-containing substances
* Received a botox injection 4 months prior to study
* Received an investigational drug within 30 days
* Previously treated with 4-aminopyridine (4-AP)
* Not on stable medication dosing in 3 weeks prior to study
* Abnormal ECG or laboratory value at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2002-06; Primary Completion 2003-11 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blight, MD, Study Director — Acorda Therapeutics
Locations (30):
- United States (27):
  - UAB School of Medicine, 190 Spain Rehab Center, Birmingham, Alabama
  - Long Beach VA Medical Center, Long Beach, California
  - University of California, Davis, Sacramento, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Craig Hospital, Englewood, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Hines VA Hospital, Hines, Illinois
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Rehabilitation Institute of Michigan, Detroit, Michigan
  - Minneapolis VA Hospital, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - University of Rochester/Strong Memorial Hospital, Rochester, New York
  - SUNY Upstate Clinical Trials Office, Syracuse, New York
  - Helen Hayes Hospital, West Haverstraw, New York
  - Charlotte Institute of Rehabilitation, Charlotte, North Carolina
  - Coastal AHEC, Wilmington, North Carolina
  - Ohio State University, Columbus, Ohio
  - Miami Valley Hospital- Rehabilitation Institute of Medicine, Dayton, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - VA North Texas Health Care System, Dallas, Texas
  - Southwestern Medical Center at Dallas, Dallas, Texas
  - INOVA Institute of Research and Education, Falls Church, Virginia
  - Medical College of Virginia/VCU, Richmond, Virginia
  - University of Washington Medical Center, Dept. of Rehabilitation, Seattle, Washington
  - Wood VA Medical Center, Milwaukee, Wisconsin
- Canada (3):
  - Health Sciences Centre, Winnipeg, Manitoba
  - Chedoke-McMaster Hospital, Hamilton, Ontario
  - St. Mary's of the Lake Hospital, Kingston, Ontario

REFERENCES:
- See also: Related Info — http://www.acorda.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The randomization schedule was created prior to the start of the study, and was blocked and stratified by site and by concomitant anti-spasmodic medication status to ensure treatment balance between patients who were treated with anti-spasmodic medications upon entry into the study and those who were not.
Pre-assignment Details: Investigational drug assignments were communicated through an Interactive Voice Response System (IVRS).
Groups:
- Fampridine-SR 50mg/Day: Fampridine-SR : 25mg bid (twice daily)
- Placebo: Placebo : Placebo
Period: Overall Study
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Started | 104 | 100
Intent to Treat (ITT) Population | 103 | 100
Safety Population | 103 | 100
Efficacy Population | 89 | 93
Completed | 78 | 88
Not Completed | 26 | 12
Not completed — Adverse Event | 12 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Population: 104 patients randomized to Fampridine-SR 50mg/day 100 patients randomized to Placebo. Total patients randomized = 204.
  Overall, 203 (99.5%) patients were included in the ITT population, 182 (89.2%) in the Efficacy population and 203 (99.5%) in the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fampridine-SR 50mg/Day | Placebo | Total
Number analyzed (Participants) | 103 | 100 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (11.79) | 40.5 (12.25) | 40.9 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 86 | 86 | 172
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 92 | 87 | 179
  Black or African American | 8 | 10 | 18
  Asian/Pacific Islander | 1 | 0 | 1
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Change From Baseline in Ashworth Score Evaluating Spasticity
Description: The Ashworth evaluates the functioning of two lower extremity muscle groups, the hamstring and quadriceps muscles, while in the supine position. The test measures extension of the right and left hamstring muscle and flexion of the right and left quadriceps muscle using the following 5-point grading scale:
  1=no increased tone; 2=slight increase in tone, giving a "catch" when the affected part is moved in flexion or extension; 3=more marked increase in tone, but affected part is easily flexed; 4=considerable increase in tone, passive movement is difficult; 5=affected part is rigid in flexion and extension.
  The Ashworth Score was determined by adding all individual scores for each muscle group and dividing by four. Higher Ashworth Scores indicated greater spasticity.
Time Frame: Baseline (visits 2,3) average score days 7,14 and double-blind treatment period (visits 4-7) average score days 28-98
Population: Intent to Treat (ITT) Population. Number of participants analyzed is number of patients with available data at both baseline and double-blind treatment period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.28 (0.046) | -0.16 (0.047)

2. Primary Outcome: Double-blind Change From Baseline in Mean Subject's Global Impression (SGI) Scores
Description: The SGI is a 7-unit ordinal scale used by the subject to evaluate the effects of study medication on his/her quality of life during the preceding week, with higher scores denoting greater satisfaction. A positive change score in SGI signifies improved outcome.
  The questionnaire consisted of one question (How do you feel about the effects of the investigational drug over the past 7 days?). The answer was based on a numerical rating scale where 1=terrible; 2=unhappy; 3=mostly dissatisfied; 4=neutral/mixed; 5=mostly satisfied; 6=pleased; 7=delighted.
Time Frame: Baseline (visits 2,3) average score days 7,14 and double-blind treatment period (visits 4-7) average score days 28-98
Population: ITT population. Number of participants analyzed is number of patients with available data at both baseline and double-blind treatment period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.0 (0.07) | 0.1 (0.08)

3. Secondary Outcome: Double-blind Change From Baseline in Mean Spasm Frequency/Severity Scores
Description: The Spasm Frequency score is the average rating by the clinician of the left and right arm(s) and leg(s), each evaluated on a 4-point scale (from 0=no spasms to 4=spontaneous spasms occurring more than ten times per hour), with higher scores denoting a greater degree of muscle spasms.
  The Spasm Severity score is the average rating of the left and right arm(s) and leg(s), each evaluated on a three-point scale (mild, moderate, or severe) as rated by the clinician on the basis of patient self-report.
  On both, a negative change in score signifies improvement in muscle spasms. The average Spasm Frequency/Spasm Severity Score was calculated as the average of the left and right non-missing scores.
Time Frame: Baseline (visits 2,3) average score days 7,14 and double-blind treatment period (visits 4-7) average score days 28-98
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale
  Arm Spasm Frequency | -0.13 (0.051) | 0.02 (0.053)
  Leg Spasm Frequency | -0.12 (0.051) | -0.10 (0.052)
  Arm Spasm Severity | -0.09 (0.034) | -0.02 (0.035)
  Leg Spasm Severity | -0.14 (0.040) | -0.07 (0.041)

4. Secondary Outcome: Double-blind Change From Baseline in Mean Clinician's Global Impression (CGI) Scores
Description: The supervising clinician rated the patient's neurological condition following treatment as compared to the screening visit on a seven-point scale (from 1=very much improved to 7=very much worse). The assessment was based on the clinician's overall impression of the patient's neurological status (specifically bowel, bladder, and sexual function; spasticity; and other neurological functions) and general state of health related to his or her participation in the study. Negative change scores indicated a change for the better.
Time Frame: Baseline (visits 2,3) average of days 7-14 and double-blind treatment period (visits 4-7) average of days 28-98)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.2 (0.06) | -0.2 (0.06)

5. Secondary Outcome: Stable-dose Change From Baseline in Mean American Spinal Injury Association(ASIA) Total Motor Score
Description: Ten key muscle groups for the right and left sides were rated on a 0 (absent) to 5 (normal) scale, with a possible total score of 100. Higher positive change scores indicate improved motor function.
Time Frame: Baseline (visits 2,3) average score days 7,14 and stable-dose treatment period (visits 5-7) average score days 56-98
Population: ITT Population. Number of participants analyzed is number of patients with available data at both baseline and stable-blind treatment period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 87 | 92
units on a scale | 0.4 (0.51) | 0.7 (0.49)

6. Secondary Outcome: Change From Baseline in Mean International Index of Erectile Function (IIEF) Score
Description: Male patients were asked to complete the IIEF questionnaire on sexual function. The IIEF is a brief, reliable, and valid self-administered questionnaire of 15 questions (items) that were categorized into five domains: Erectile Function (EF) scores: 0-6 Severe dysfunction, 7-12 Moderate dysfunction, 13-18 Mild to moderate dysfunction, 19-24 Mild dysfunction, 25-30 No dysfunction. Orgasmic Function (OF) score range: 0-2 Severe dysfunction to 9-10 No dysfunction, Sexual Desire (SD) score range: 0-2 Severe dysfunction to 9-10 No dysfunction, Intercourse Satisfaction (IS) score range: 0-3 Severe dysfunction to 13-15 No dysfunction, and Overall Satisfaction (OS) score range: 0-2 Severe dysfunction to 9-10 No dysfunction.
  Domain scores were derived by summing the individual items within a given domain. Final scale ranges from 0 (negative) to 5 (positive). A positive change in IIEF domain scores signifies improvement.
Time Frame: Baseline (visit 1) average score obtained at day 1 and stable treatment period (visit 7) average score day 98
Population: ITT Population. N = number of participants analyzed with available data at both baseline and stable treatment period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 65 | 77
units on a scale
  EF (Fampridine-SR Number (N) =65, Placebo N=77) | 0.8 (1.09) | 1.6 (1.01)
  OF (Fampridine-SR N=64, Placebo N=76) | 0.3 (0.36) | 0.0 (0.33)
  SD (Fampridine-SR N=64, Placebo N=75) | -0.0 (0.23) | 0.0 (0.21)
  IS (Fampridine-SR N=64, N=76) | 0.4 (0.55) | 0.4 (0.50)
  OS (Fampridine-SR N=51, Placebo N=66) | 0.4 (0.27) | 0.3 (0.24)

7. Secondary Outcome: Change From Baseline in Mean Female Sexual Function Index (FSFI) Scores
Description: The FSFI is a brief, reliable, and valid self-administered questionnaire of 19 questions (items). It contains six domains: Desire (2 items score range: 1 Very low or none at all to 5 Very high), Arousal (4 items score range: 0 No sexual activity to 5 Almost always or always), Lubrication (4 items score range: 0 No sexual activity to 5 Almost always or always), Orgasm (3 items score range: 0 No sexual activity to 5 Almost always or always), Satisfaction (3 items score range: 0 No sexual activity to 5 Very satisfied) and Pain (3 items score range: 0 Did not attempt intercourse to 5 Almost never or never).
  A positive change signifies improvement.
Time Frame: Baseline (visit 1) average score obtained at day 1 and stable treatment period (visits 4-7) average score days 28-98
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale
  Desire | 0.7 (0.26) | 0.2 (0.28)
  Arousal | 0.6 (0.37) | 0.2 (0.40)
  Lubrication | 0.7 (0.45) | -0.2 (0.48)
  Orgasm | 0.2 (0.18) | 0.4 (0.19)
  Satisfaction (Fampridine-SR N=13, Placebo N=12) | 0.4 (0.25) | 0.3 (0.26)
  Pain | 0.7 (0.47) | -0.1 (0.50)

8. Secondary Outcome: Adjusted Mean Change in Subject Bladder/Bowel Function Diary Scores
Description: Bowel/bladder questions pertaining to the average number of times per day the patient experienced accidental urination/leakage and the average number of bowel movements per day were asked of all patients daily.
  A negative change in patient bladder/bowel function diary score signifies improvement.
Time Frame: Baseline (visit 1) average score obtained at day 1 and double-blind treatment period (visits 4-7) average score days 28-98
Population: as for outcome 2
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 103 | 99
episodes
  Number of Accidental Urination or Leakage | -0.2 (0.20) | -0.2 (0.21)
  Number of Bowel Movements | 0.1 (0.03) | -0.0 (0.03)

9. Secondary Outcome: Adjusted Mean Change in Subject Bowel Function Diary Scores
Description: Bowel questions pertaining to the average number of minutes per day spent on bowel routine were asked of all patients daily.
  A negative change in patient bowel function diary score signifies improvement.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 103 | 99
minutes | -0.7 (0.90) | 0.3 (0.93)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAE) include AEs with date of onset (or worsening) on or after the start of treatment and no more than 14 days after the last dose of investigational drug.
Description: Adverse events were recorded at every study visit. Results are presented for the Safety population defined as all randomized patients who received at least one dose of study treatment.
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 8/103 | 9/100
Other Adverse Events (participants affected / at risk) | 24/103 | 17/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR 50mg/Day (N=103) | Placebo (N=100)
Accidental Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypothermia (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Psychiatric disorders) | 0 (0) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Myocardial Infarct (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysautonomia (Nervous system disorders) | 1 (1) | 3 (3)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Speech Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR 50mg/Day (N=103) | Placebo (N=100)
Hypertonia (Psychiatric disorders) | 24 (32) | 17 (21)
Urinary Tract Infection (Infections and infestations) | 22 (33) | 15 (22)
Pain (General disorders) | 19 (23) | 14 (15)
Constipation (Renal and urinary disorders) | 19 (23) | 10 (12)
Paresthesia (Nervous system disorders) | 18 (25) | 9 (11)
Insomnia (Psychiatric disorders) | 16 (17) | 6 (8)
Headache (Nervous system disorders) | 15 (20) | 8 (11)
Dizziness (Vascular disorders) | 12 (12) | 1 (1)
Infection (Infections and infestations) | 11 (12) | 15 (15)
Abdominal Pain (Gastrointestinal disorders) | 10 (11) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (16) | 3 (6)
Accidental Injury (Injury, poisoning and procedural complications) | 9 (10) | 16 (22)
Nausea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Peripheral Edema (General disorders) | 7 (8) | 9 (10)
Fever (General disorders) | 6 (9) | 5 (6)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Flu Syndrome (Infections and infestations) | 5 (5) | 0 (0)
Migraine (Nervous system disorders) | 5 (7) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 5 (10)
Ecchymosis (Vascular disorders) | 5 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Nervousness (Psychiatric disorders) | 5 (6) | 2 (2)
Cough Increased (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 7 (7)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (6)
Sweating (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1)
Rhinitis (Infections and infestations) | 4 (5) | 4 (4)
Urinary Frequency (Renal and urinary disorders) | 4 (4) | 4 (5)
Urinary Incontinence (Renal and urinary disorders) | 4 (4) | 4 (4)
Asthenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (8)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck Rigidity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (7) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Leukocvtosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Abnormal Dreams (Psychiatric disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Dysautonomia (Nervous system disorders) | 3 (3) | 5 (5)
Vasodilatation (Vascular disorders) | 3 (4) | 1 (1)
Dyspnea (Cardiac disorders) | 3 (4) | 1 (1)
Cystitis (Renal and urinary disorders) | 3 (4) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (3) | 3 (6)
Urine Abnormality (Renal and urinary disorders) | 3 (3) | 2 (2)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (9)
Neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Fungal Dermatitis (Infections and infestations) | 2 (2) | 2 (2)
Amblyopia (Eye disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.